CLINICAL TRIAL: NCT06987019
Title: Reliability and Validity of Continuous Inter-Limb Stability in Veterans With Lower Limb Loss
Brief Title: Reliability and Validity of Continuous Inter-limb Stability
Acronym: CS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: A5147-P
Record Dates: First submitted 2025-04-11; First posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Amputation, Lower Limb
Keywords: Transtibial amputation; Gait evaluation
MeSH Terms: interventions — Wearable Electronic Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Reliability and Validity (Experimental): Reliability and Validity of Inter-limb Stability using 3D motion capture, functional outcome measures, and wearable devices
  Interventions: Other: 3D motion capture, wearable devices, and functional outcome measures

INTERVENTIONS:
Other: 3D motion capture, wearable devices, and functional outcome measures — Gait evaluation, Hill and Stair Assessment Indices, 6 minute walk test, AMPPro, Timed Up and Go

SUMMARY:
To date, there is no valid and reliable measure of continuous inter-limb stability available to healthcare teams treating people with lower limb loss. Determining these characteristics of this parameter for this population is important because superior stability has been linked to increased physical activity and strength in similar populations, making it a potential vital contributor to mobility improvement of Veterans with limb loss. It is also crucial that healthcare providers can easily measure continuous stability in the clinic instead of relying on expensive laboratory equipment. The overall goals of this study are to determine the reliability and validity of continuous inter-limb stability of Veterans with lower limb loss and determine if this parameter can be captured using accessible wearable technology. Consequently, clinicians can improve continuous stability through proper rehabilitation to positively impact the functional mobility and overall quality of life of Veterans with lower limb loss.

DETAILED DESCRIPTION:
There is currently no valid or reliable biomechanical variable available to objectively measure the continuous stability of Veterans with lower limb loss. However, continuous inter-limb stability represents a potential target to improve whole-body dynamics, as it is an important measure of functional mobility in individuals with lower limb loss. Determining the reliability and validity of this measure is critical for limb loss care teams since these features are fundamental to interpretability and assessment of this parameter. Unlike traditional clinical assessments of stability that focus on the time of task execution, Relative Phase (RP) analysis, which is a novel methodology that can be used to evaluate continuous stability, uses both space and time within one outcome variable. While previous literature supports the use of continuous stability for mobility challenged populations, such as individuals with limb loss, it has yet to be shown reliable and valid for such populations. Therefore, the first aim of this study is to identify the reliability and validity of continuous inter-limb stability in individuals with transtibial limb loss (TLL) using RP analysis. For this parameter to be used clinically, it is vital to provide rehabilitation specialists the ability to assess continuous stability within the clinical setting. To date, this factor of functional mobility has only been evaluated using 3-dimensional (3-D) motion capture, which is costly and inaccessible to most rehabilitation clinics. Therefore, the second aim of this study is to identify the strength of the association between wearable technology (using inertial measurement units) and 3-D motion capture system for evaluation of continuous interlimb stability of individuals with TLL. The central hypothesis is that continuous stability evaluated using RP analysis will be a reliable and valid measure of functional mobility for Veterans with TLL and that data captured via wearable technology will be strongly associated with 3-D analysis. Twenty Veterans with TLL will be recruited and enrolled via the Prosthetic or Physical Medicine Departments at Veterans Affairs New York Harbor Healthcare System, where all data collection will occur. To measure test re-test reliability, participants will undergo 3 sessions of 3-D gait analysis while walking at a moderate speed (1.3m/s) until 15 walking cycles are captured, with 1 day between sessions. RP analysis will be used to identify the continuous inter-limb stability of gait patterns. Participants will be fit with wearable technology and data will be collected concurrently. To measure convergent validity, participants will perform functional outcome measures including the Timed Up and Go test, 6 Minute Walk Test, Hill and Stair Assessment Indexes, and Amputee Mobility Predictor. Data from 40 participants are required to appropriately power the analysis of convergent validity. To achieve this power, data from 20 participants collected during a previously funded Department of Defense study will be leveraged and added to the data of the 20 participants collected during the proposed study. This is possible due to identical data collection techniques in both studies. To assess the level of agreement between the data obtained from the 3 sessions, Intraclass Correlation Coefficients will be calculated for each variable, in addition to Cohen's kappa statistics and Pearson correlation coefficients. To assess convergent validity, Pearson and Spearman rank correlation coefficients will quantify the strength and direction of the relationships between the outcome measures and continuous stability. Substantiating the use of continuous stability in Veterans with TLL will afford healthcare providers information necessary to accurately detect and appropriately address stability deficiencies, which is critical since superior stability is linked to increased physical activity leading to an enhanced overall quality of life of Veterans with limb loss. Verifying the reliability and validity of this parameter will lead to its confident application for future studies focused on effectiveness, optimization, and rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* any individual with unilateral transtibial limb loss
* a well-fitting prosthesis (as determined by a board-certified prosthetist through standardized prosthetic guidelines) for a minimum of one month
* able to achieve a "Level 6 - Modified Independence" score on the Functional Independence Measure (FIM) for 2 mobility items (locomotion and transfers)

Exclusion Criteria:

* Individuals with active wounds/ulcers or significant musculoskeletal comorbidities on their intact limb that would impair ability to participate in biomechanical evaluations
* any comorbidity that results in rapid limb volume changes (i.e., end stage renal disease with dialysis)
* a poorly fitting socket
* cognitive deficit(s) or mental pathology (e.g., dementia, amnesia) that would prevent the participant from understanding and following directions and limit the participant's ability to participate fully in the study
* women who are pregnant or who plan to become pregnant during their participation in study activities
* FIM scores less than Level 6 for locomotion and transfers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Reliability of Continuous Inter-limb Stability | 3 times at visits 2-4 (once per visit) (will occur within 1 week)
  Reliability will be evaluated using Deviation Phase using Relative Phase Analysis. Deviation Phase measures the continuous stability of two oscillating segments throughout a cyclical movement. Relative Phase Analysis is a dynamical systems based methodology that is used to calculated the continuous stability of a movement, such as walking. Deviation Phase ranges from 0-180 degrees, with a lower value indicating better organization of the neuromuscular system.
Convergent Validity of Continuous Inter-limb Stability - TUG | Once at visit 2 of 4 (Baseline)
  The TUG measures physical mobility in individuals with lower limb loss. This measures the time it takes for an individual to stand up from a standard arm chair, walk a distance of 10 feet, turn, walk back to the chair, and sit down. This is measured in time (seconds).
Convergent Validity of Continuous Inter-limb Stability - 6MWT | Once at visit 2 of 4 (Baseline)
  The 6MWT measure function and endurance. This test measures the distance an individual can walk in 6 minutes without help. This is measured in meters.
Convergent Validity of Continuous Inter-limb Stability - SAI | Once at visit 2 of 4 (Baseline)
  The SAI is a graded qualitative scale on how an individual with lower limb amputation negotiates up and down a staircase. This is measured on a scale of 0-13.
Convergent Validity of Continuous Inter-limb Stability - HAI | Once at visit 2 of 4 (Baseline)
  The HAI is a graded qualitative scale on how an individual with lower limb amputation negotiates up and down a ramp. This is measured on a scale from 0-11.
Convergent Validity of Continuous Inter-limb Stability - AMPPro | Once at visit 2 of 4 (Baseline)
  The AMPPro is a 21 item instrument designed to measure basic prosthetic mobility of individuals with lower extremity amputation. This is scored from 0-47.

SECONDARY OUTCOMES:
Strength of association between wearable technology and 3D motion capture to measure inter-limb stability | 3 times at visits 2-4 (once per visit) (will occur within 1 week)
  Correlation between IMUs and Motion Capture. Xsens IMUs consist of 3 measurement sensor categories: accelerometer, gyroscope, and magnetometer, with measurements of all 3 axes. The accelerometer provides linear acceleration of the deice. The Gyroscope measures the angular rate and is then integrated to determine the angle of the sensor. The magnetometer detects magnetic field, use as an external reference frame. The 3 signals combine to produce a sensor coordinate system, while the signal variety eliminates drift effects commonly found in gyroscopic measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Alexis Sidiropoulos, PhD, Principal Investigator — VA NY Harbor Healthcare System, New York, NY
Locations (1):
- VA NY Harbor Healthcare System, New York, NY, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data will be stored in a curated data repository that makes the data underlying scientific publications discoverable, freely usable, and citable, while promoting openly available research integrated with scholarly literature.
Time Frame: After study completion